CLINICAL TRIAL: NCT02806986
Title: A Multi-Center, Open-Label, Single-Arm Trial to Evaluate Efficacy, Pharmacokinetics, and Safety and Tolerability of IGSC 20% in Subjects With Primary Immunodeficiency
Brief Title: Efficacy, Pharmacokinetics, Safety, and Tolerability of IGSC 20% in Subjects With Primary Immunodeficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTI1503; 2015-003290-15 (EudraCT Number)
Record Dates: First submitted 2016-06-03; First posted 2016-06-21 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Caprylates; Chromatography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IGSC 20% (Experimental): 13 doses of IGSC 20% in Treatment Stage 1 and 39 doses of IGSC 20% in Treatment Stage 2 for a total of 52 doses if IGSC 20%
  Interventions: Biological: IGSC 20%

INTERVENTIONS:
Biological: IGSC 20% — Weekly administration of IGSC 20% via intravenous infusion
  Other Names: Immune Globulin Subcutaneous (Human), 20% Caprylate/Chromatography

SUMMARY:
Approximately 60 subjects will be enrolled in order to have approximately 20 adult subjects and 20 pediatric subjects treated with subcutaneously administered Immune Globulin Subcutaneous (Human), 20% Caprylate/Chromatography Purified (IGSC 20%) who complete the entire study. This study will include 3 study stages: Screening/Previous Regimen Phase, IGSC 20% Treatment Stage 1 (13 IGSC 20% weekly doses), and IGSC 20% Treatment Stage 2 (39 IGSC 20% weekly doses). A total of 52 doses of IGSC 20% will be administered with a final follow-up visit 1 week after the last dose at Week 53. Subjects/caregivers will be trained on self-administration of IGSC 20% by the clinical site personnel.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, single-arm, efficacy, PK, safety and tolerability study of IGSC 20% in subjects with PI. Approximately 60 subjects will be enrolled in order to have approximately 20 adult subjects and 20 pediatric subjects treated with subcutaneously administered IGSC 20% who complete the entire study.

This study will include 3 study stages: Screening/Previous Regimen Phase, IGSC 20% Treatment Stage 1 (13 IGSC 20% weekly doses), and IGSC 20% Treatment Stage 2 (39 IGSC 20% weekly doses).

Previous Regimen Phase: Subjects will be infused with their current ongoing ("previous regimen") intravenous immune globulin/subcutaneous immune globulin (IVIG/SCIG) regimen (pIV/pSC) in the clinic to obtain 2 trough immunoglobulin G (IgG) levels (obtained prior to each pIV/pSC infusion) on each subject's "previous regimen".

20% IGSC Treatment Stage 1: The first dose of IGSC 20% will be administered at the clinical site immediately after Baseline assessments are complete (SC#1). All subjects will receive 13 IGSC 20% infusions at weekly intervals. IgG trough blood levels will be measured at all (except SC#3) study visits All other doses of IGSC 20% may be infused at home (once properly trained) or in the clinic. The Treatment Stage 1 dose will continue into IGSC 20% Treatment Stage 2.

IGSC 20% Treatment Stage 2: The IGSC 20% dose (mg/kg) will remain constant with no dose adjustment permitted in this phase, unless it is absolutely medically necessary. While all subjects will have a SC#17 clinic visit and standard assessments, serial pharmacokinetics (PK) sampling will only be performed in a subset of adult subjects:

ELIGIBILITY:
Inclusion Criteria:

* Pre-existing diagnosis of PI with features of hypogammaglobulinemia requiring IgG replacement therapy
* No serious bacterial infection within the 3 months prior to Screening and has no serious bacterial infections (SBIs) up to the time of the Baseline Visit
* Currently on IgG replacement therapy (stable regimen [dose and dosing interval] via IV or SC infusion) for ≥ 3 consecutive months at a dosage of at least 200 mg/kg per infusion
* Documented (within previous 3 months) of an IgG trough level of ≥ 500 mg/dL on current IgG replacement therapy regimen
* Screening/pre-Baseline trough IgG levels must be ≥ 500 mg/dL.

Exclusion Criteria:

* Known serious adverse reaction to immunoglobulin or any severe anaphylactic reaction to blood or any blood-derived product
* History of blistering skin disease, clinically significant thrombocytopenia, bleeding disorder, diffuse rash, recurrent skin infections, or other disorders where SC therapy would be contraindicated during the study
* Isolated IgG subclass deficiency, isolated specific antibody deficiency disorder, or transient hypogammaglobulinemia of infancy
* Nephrotic syndrome, and/or a history of acute renal failure, and/or severe renal impairment, and/or is on dialysis
* Known previous infection with or clinical signs and symptoms consistent with current hepatitis B virus or hepatitis C virus infection
* History of (year prior to Screening or 2 episodes in lifetime) or current diagnosis of deep venous thrombosis or thromboembolism (e.g., myocardial infarction, cerebrovascular accident, or transient ischemic attack)
* Acquired medical condition known to cause secondary immune deficiency, such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, chronic or recurrent neutropenia (absolute neutrophil count less than 1000/μL [1.0 x 10^9/L]), or human immunodeficiency virus infection/acquired immune deficiency syndrome
* HIV positive by nucleic acid amplification technology based on a Screening blood sample
* Uncontrolled arterial hypertension (adult subjects: systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg)
* Receiving any of the following medications: (a) immunosuppressants including chemotherapeutic agents, (b) immunomodulators, (c) long-term systemic corticosteroids defined as daily dose > 1 mg of prednisone equivalent/kg/day for > 30 days Note: Intermittent courses of corticosteroids of not more than 10 days would not exclude a subject. Inhaled or topical corticosteroids are allowed.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- Australia (2):
  - Wesley Medical Research, Auchenflower
  - Royal Melbourne Hospital, Parkville
- University Hospital, Hradec Králové, Czechia
- CHU de Montpellier, Montpellier, France
- Germany (5):
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Children's Hospital at Municipal Hospital St. Georg, Leipzig
  - University Hospital of Mainz, Mainz
  - Asklepios Klinik Sankt Augustin, Sankt Augustin
- Hungary (2):
  - United St Istvan and St Laszlo Hospital, Budapest
  - Josa Andras County Hospital, Nyiregyháza
- The Children's Memorial Health Institute, Warsaw, Poland
- Spain (7):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitari Sant Joan de Déu, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Clinico San Carlos, Madrid
  - Hospital 12 Octubre, Madrid
  - Hospital Virgen del Rocio, Seville
- Stockholm, Stockholm, Sweden
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge
  - St Bartholomew's Hospital, London
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with primary immunodeficiency (PI) requiring IgG replacement were enrolled. Study has 3 stages: Screening/Previous Regimen Phase, Treatment Stage 1 and 2. Total 62 participants entered Previous Regimen Phase, of which 61 entered in Treatment Stage 1 to receive IGSC 20%. Study was conducted in 8 countries from June 2016 to May 2019.
Pre-assignment Details: Participants had no SBI within last 3 months prior to screening and were on immunoglobulin G (IgG) replacement therapy (stable regimen via intravenous [IV] or subcutaneous [SC] infusion) for ≥3 consecutive months prior to screening. Participants receiving IVIG prior to study entry must have received a dosage of ≥200 mg/kg per infusion.
Groups:
- IGSC 20%: Following the previous regimen phase (screening), participants were enrolled to receive 13 immune globulin subcutaneous (human), 20% caprylate/chromatography purified (IGSC 20%) infusions at weekly intervals from baseline (Week 1) up to Week 13 in treatment stage 1. Participants were infused with IGSC 20% at a 1:1 dose-equivalent regimen from their previous regimen (or a minimum IGSC 20% dose of 100 milligram per kilogram per week (mg/kg/week) if the derived 1:1 dose from the previous regimen was lower) and followed by 39 IGSC 20% infusions at weekly intervals from Week 14 up to Week 52 in treatment stage 2. Dose adjustments were permitted per the study protocol and at the Investigator's discretion in the treatment stage 1. However, dose remained constant in treatment stage 2 unless it was absolutely medically necessary to change the dose, and such change required prior consultation with the Sponsor's Medical Monitor. A final follow-up visit occurred at Week 53.
Period: Treatment Stage 1
Arm/Group | IGSC 20%
Started | 61
Completed | 60
Not Completed | 1
Not completed — Adverse Event | 1
Period: Treatment Stage 2
Arm/Group | IGSC 20%
Started | 60
Completed | 55
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The efficacy evaluable population included all participants who received at least 1 dose of IGSC 20%.
Groups:
- IGSC 20%: Following the previous regimen phase (screening), participants were enrolled to receive 13 IGSC 20% infusions at weekly intervals from baseline (Week 1) up to Week 13 in treatment stage 1. Participants were infused with IGSC 20% at a 1:1 dose-equivalent regimen from their previous regimen (or a minimum IGSC 20% dose of 100 mg/kg/week if the derived 1:1 dose from the previous regimen was lower) and followed by 39 IGSC 20% infusions at weekly intervals from Week 14 up to Week 52 in treatment stage 2. Dose adjustments were permitted per the study protocol and at the Investigator's discretion in the treatment stage 1. However, dose remained constant in treatment stage 2 unless it was absolutely medically necessary to change the dose, and such change required prior consultation with the Sponsor's Medical Monitor. A final follow-up visit occurred at Week 53.
Arm/Group | IGSC 20%
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (19.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 57
  American Indian or Alaska Native | 2
  Unknown | 2
Subject Entry Status [Count of Participants; unit: Participants]
  Entered on intravenous immune globulin (IVIG) | 40
  Entered on subcutaneous immune globulin (SCIG) | 21

OUTCOME MEASURES:

1. Primary Outcome: Rate of Serious Bacterial Infection (SBI) Per Participant Per Year
Description: The rate of SBI events per participant per year during IGSC 20% treatment was calculated as the total number of SBI events divided by the total duration of exposure in years across all participants. The 2-sided 98% confidence interval (CI) was determined from a generalized linear model for poisson regression for the log-transformed number of events with log-transformed duration of exposure in years as an offset variable.
Time Frame: IGSC 20% Treatment Stage 1: Week 1 to 13; IGSC 20% Treatment Stage 2: Week 14 to 53; IGSC 20% Overall: Week 1 to 53
Population: Analysis was performed on the efficacy evaluable population which included all participants who received at least 1 dose of IGSC 20%.
Measure: Number (98% Confidence Interval); unit: Rate of events per participant per year
Groups:
- IGSC 20% Treatment Stage 1: Following previous regimen phase (screening), participants were enrolled to receive 13 IGSC 20% infusions at weekly intervals from baseline (Week 1) up to Week 13. Participants were infused with IGSC 20% at a 1:1 dose-equivalent regimen from their previous regimen (or a minimum IGSC 20% dose of 100 mg/kg/week if the derived 1:1 dose from the previous regimen was lower). Dose adjustments were permitted in this phase per the study protocol and at the Investigator's discretion.
- IGSC 20% Treatment Stage 2: Following treatment stage 1, participants received 39 IGSC 20% infusions at weekly intervals from Week 14 up to Week 52. The IGSC 20% dose (mg/kg) remained constant with no dose adjustment permitted in this phase, unless it was absolutely medically necessary to change the dose, and such change required prior consultation with the Sponsor's Medical Monitor. A final follow-up visit occurred at Week 53.
- IGSC 20% Overall: Following previous regimen phase (screening), participants were enrolled to receive 13 IGSC 20% infusions at weekly intervals from baseline (Week 1) up to Week 13 in treatment stage 1. Participants were infused with IGSC 20% at a 1:1 dose-equivalent regimen from their previous regimen (or a minimum IGSC 20% dose of 100 mg/kg/week if the derived 1:1 dose from the previous regimen was lower) and followed by 39 IGSC 20% infusions at weekly intervals from Week 14 up to Week 52 in treatment stage 2. Dose adjustments were permitted per the study protocol and the at Investigator's discretion in the treatment stage 1. However, dose remained constant in treatment stage 2 unless it was absolutely medically necessary to change the dose, and such change required prior consultation with the Sponsor's Medical Monitor. A final follow-up visit occurred at Week 53.
Arm/Group | IGSC 20% Treatment Stage 1 | IGSC 20% Treatment Stage 2 | IGSC 20% Overall
Number analyzed (Participants) | 61 | 60 | 61
Rate of events per participant per year | 0 [NA to NA] — Here NA signifies that 98% CI was not estimable due to zero number of events. | 0.023 [0.008 to 0.049] | 0.017 [0.006 to 0.036]

2. Secondary Outcome: Mean Trough Total IgG Concentration
Description: Mean trough total IgG concentration during the previous regimen phase was calculated as the average of the trough concentrations at the previous IVIG (pIV)#1 and pIV#2 visits for participants entering the study on a previous IVIG regimen, or at the previous subcutaneous immune globulin (SCIG) (pSC)#1 and baseline/SC#1 visits for participants entering the study on a previous SCIG regimen. Mean trough total IgG concentration during the IGSC 20% phase was calculated as the average of all steady state trough concentrations measured during the IGSC 20% treatment stage 2 at the visits corresponding to Weeks 17, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52 and 53.
Time Frame: Previous Regimen Phase: 2 timepoints pre-dose of pIV or pSC between Screening and Baseline (up to 8 weeks). IGSC 20% Phase: Pre-dose of IGSC 20% at Baseline (Week 1), Weeks 2, 5, 9, 13, 17, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52, and at Week 53
Population: Analysis was performed on the IgG population which consisted of all participants who received any amount of IGSC 20% and had total IgG concentration data to facilitate the comparison of mean trough IgG concentration during the IGSC 20% phase versus the pre-treatment phase.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Groups:
- Previous Regimen: Participants were required to attend the clinic for infusion with their previous ongoing ("previous regimen") IVIG/SCIG regimen (pIV/pSC) to obtain 2 trough IgG levels (obtained prior to each pIV/pSC infusion) on each participant's "previous regimen". Trough levels for total IgG determined during the Previous Regimen Phase were used to confirm final eligibility for participants entering the study to receive treatment with IGSC 20% (must be ≥500 milligrams per deciliter [mg/dL]).
Arm/Group | IGSC 20% Overall | Previous Regimen
Number analyzed (Participants) | 59 | 59
milligram per deciliter (mg/dL) | 947.64 (150.262) | 891.37 (165.943)

3. Secondary Outcome: Rate of Infection of Any Kind Per Participant Per Year
Description: The total number of infections of any kind (serious/non-serious including acute sinusitis, exacerbation of chronic sinusitis, acute otitis media, pneumonia, acute bronchitis, infectious diarrhea, etc.) as determined by the investigator were evaluated. The rate of infection events per participant per year during IGSC 20% treatment was calculated as the total number of infection events divided by the total duration of exposure in years across all participants. The 2-sided 95% CI was determined from a generalized linear model for poisson regression for the log-transformed number of events with log-transformed duration of exposure in years as an offset variable.
Time Frame: IGSC 20% Treatment Stage 1: Week 1 to 13; IGSC 20% Treatment Stage 2: Week 14 to 53; IGSC 20% Overall: Week 1 to 53
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Rate of events per participant per year
Arm/Group | IGSC 20% Treatment Stage 1 | IGSC 20% Treatment Stage 2 | IGSC 20% Overall
Number analyzed (Participants) | 61 | 60 | 61
Rate of events per participant per year | 2.524 [1.720 to 3.547] | 2.353 [1.736 to 3.102] | 2.397 [1.824 to 3.079]

4. Secondary Outcome: Rate of Days on Antibiotics Per Participants Per Year
Description: The rate of days on antibiotics per participants per year during IGSC 20% treatment was calculated as the total number of days on antibiotic divided by the total duration of exposure in years across all participants. The 2-sided 95% CI was determined from a generalized linear model for poisson regression for the log transformed number of days with log-transformed duration of exposure in years as an offset variable.
Time Frame: IGSC 20% Treatment Stage 1: Week 1 to 13; IGSC 20% Treatment Stage 2: Week 14 to 53; IGSC 20% Overall: Week 1 to 53
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Rate of days per participant per year
Arm/Group | IGSC 20% Treatment Stage 1 | IGSC 20% Treatment Stage 2 | IGSC 20% Overall
Number analyzed (Participants) | 61 | 60 | 61
Rate of days per participant per year
  Prophylactic Antibiotic | 43.240 [24.786 to 69.152] | 44.846 [26.197 to 70.755] | 44.432 [26.351 to 69.339]
  Therapeutic Antibiotics | 13.085 [7.777 to 20.387] | 7.451 [4.843 to 10.861] | 8.904 [5.949 to 12.705]

5. Secondary Outcome: Rate of Hospitalization Due to Infection Per Participants Per Year
Description: The rate of hospitalization due to infection events per participant per year during IGSC 20% treatment was calculated as the total number of hospitalization due to infection events divided by the total duration of exposure in years across all participants. The 2-sided 95% CI was determined from a generalized linear model for poisson regression for the log-transformed number of events with log-transformed duration of exposure in years as an offset variable.
Time Frame: IGSC 20% Treatment Stage 1: Week 1 to 13; IGSC 20% Treatment Stage 2: Week 14 to 53; IGSC 20% Overall: Week 1 to 53
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Rate of events per person per year
Arm/Group | IGSC 20% Treatment Stage 1 | IGSC 20% Treatment Stage 2 | IGSC 20% Overall
Number analyzed (Participants) | 61 | 60 | 61
Rate of events per person per year | 0 [NA to NA] — Here NA signifies that 95% CI was not estimable due to zero number of events. | 0.023 [0.010 to 0.044] | 0.017 [0.008 to 0.033]

6. Secondary Outcome: Rate of Days of Work/School/Daily Activities Missed Per Participants Per Year Due to Infections and Related Treatment
Description: The rate of days of work, school or daily activities missed per participant per year during IGSC 20% treatment was calculated as the total number of days of work/school/daily activities missed divided by the total duration of exposure in years across all participants. The 2-sided 95% CI was determined from a generalized linear model for poisson regression for the log-transformed number of days with log transformed duration of exposure in years as an offset variable.
Time Frame: IGSC 20% Treatment Stage 1: Week 1 to 13; IGSC 20% Treatment Stage 2: Week 14 to 53; IGSC 20% Overall: Week 1 to 53
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Rate of days missed per person per year
Arm/Group | IGSC 20% Treatment Stage 1 | IGSC 20% Treatment Stage 2 | IGSC 20% Overall
Number analyzed (Participants) | 61 | 60 | 61
Rate of days missed per person per year | 4.118 [2.270 to 6.769] | 5.283 [3.192 to 8.132] | 4.983 [3.064 to 7.572]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the beginning of treatment administration with IGSC 20% (Baseline/Week 1) until the Final Visit (Week 53). Up to 1 year overall.
Description: TEAEs are presented for the safety population which included all participants who received any amount of IGSC 20%.
Arm/Group | IGSC 20% Overall
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 7/61
Other Adverse Events (participants affected / at risk) | 49/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGSC 20% Overall (N=61)
Joint dislocation (Injury, poisoning and procedural complications) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Medical device site joint pain (General disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IGSC 20% Overall (N=61)
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Headache (Respiratory, thoracic and mediastinal disorders) | 7
Infusion site erythema (General disorders) | 10
Infusion site pruritus (General disorders) | 8
Pyrexia (General disorders) | 7
Infusion site pain (General disorders) | 5
Infusion site swelling (General disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Nasopharyngitis (Infections and infestations) | 12
Upper respiratory tract infection (Infections and infestations) | 9
Bronchitis (Infections and infestations) | 8
Rhinitis (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 7
Gastroenteritis (Infections and infestations) | 6
Lower respiratory tract infection (Infections and infestations) | 5
Influenza (Infections and infestations) | 4
Viral infection (Infections and infestations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT02806986/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT02806986/SAP_001.pdf